CLINICAL TRIAL: NCT05990166
Title: Randomised Controlled Trial to Assess the Effect of a Mineral-enriched Powder on Iron Deficiency in Women of Reproductive Age
Brief Title: Assessing the Effect of a Mineral-enriched Powder on Iron Deficiency in Women of Reproductive Age
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Carleton University (Other)
Collaborators: University of Ottawa (Other); Hopital Montfort (Other); Lucky Iron Fish Enterprise (Unknown)
Responsible Party: Principal Investigator, Kristin Connor, PhD, Associate Professor, Carleton University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LIFE2022RCT2
Record Dates: First submitted 2023-05-26; First posted 2023-08-14 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Iron Deficiency; Iron Deficiency Anaemia
Keywords: Iron deficiency; Iron deficiency anaemia; Iron fortification; Reproductive-aged women
MeSH Terms: conditions — Iron Deficiencies; Anemia, Iron-Deficiency

STUDY DESIGN:
Intervention Model Description: Double-blind randomised placebo-controlled trial
Who Masked: Participant, Investigator
Masking Description: All participants, researchers, and the study physician will be blinded to the treatment group (active intervention or placebo) to which participants have been randomised. A delegated unblinded staff member will be permitted to unblind participants for safety purposes, if requested by the principal investigators or the study physician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active intervention (Experimental): Mineral-enriched powder
  Interventions: Other: Mineral-enriched powder
- Placebo (Placebo Comparator): Placebo powder
  Interventions: Other: Placebo powder

INTERVENTIONS:
Other: Mineral-enriched powder — Mineral-enriched powder Mineral-enriched powder to allow for at-home fortification of beverages with 5 mg of ferrous iron and 10 mg of zinc sulfate monohydrate
  Arms: Active intervention
Other: Placebo powder — Placebo powder which is identical to the mineral- enriched powder, but does not contain the active ingredients (ferrous iron and zinc sulfate monohydrate)
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to determine if taking a mineral-enriched powder can raise blood iron levels compared to a placebo powder in reproductive-aged women with iron deficiency. The main questions it aims to answer are:

* Does the mineral-enriched powder raise blood iron levels compared to a placebo powder in women when it is taken every day for six months?
* How many participants still have iron deficiency after six months of taking the mineral-enriched powder compared to a placebo powder?

Participants in this clinical trial will drink the mineral-enriched powder containing ferrous iron and zinc sulphate monohydrate or a placebo powder mixed with 1 litre of water daily for six months. The placebo is a look-alike substance that does not contain active ingredients (iron and zinc). Participants will also have to:

* Complete an online "study diary" every two weeks for six months
* Provide a blood sample once a month for six months
* Attend three in-person visits with a researcher, at enrolment (baseline), midline (three months), and endline (six months)
* Complete three sets of online questionnaires (following each in-person visit)
* Complete three sets of dietary assessments (following each in-person visit)
* Provide three stool samples (following each in-person visit)

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant and non-lactating
* English speaking with the ability to give informed consent
* 18-35 years of age (inclusive)
* Women who are biologically female
* Iron deficient (SF >/=12μg/L and </=30 μg/L). Note: there is currently poor consensus on diagnostic criteria for iron deficiency based on SF concentrations. Current recommendations range from 15 μg/L to 100 μg/L.
* Hb >/=110 g/L
* Willing and able to agree to the requirements and lifestyle restrictions of this study
* Able to understand and read the questionnaires in English and carry out all study-related procedures
* Located in the greater Ottawa area and a resident of Ontario

Exclusion Criteria:

* Individuals who are lactating, pregnant, or planning to become pregnant during the study
* Individuals who are not maintaining adequate birth control measures

  * Adequate birth control measures include any option that will adequately prevent pregnancy including: contraceptives, lifestyle choices, complete abstinence, or as a result of other medical methods, procedures, or conditions
* Have a known sensitivity, intolerability, or allergy to any of the study products or their excipients
* Are using vitamin and mineral supplements containing iron and/or zinc
* SF concentrations <12 μg/L or >30 μg/L
* Having moderate or severe anaemia (Hb <109 g/L)
* Expecting to change diet and exercise regimen in the next 6 months
* Are frequent blood donors

  * Have donated blood in the last four months
  * Donate blood more than two to three times per year
* Had major surgery in the past three months
* Have planned surgery during the course of the study
* History of problematic alcohol or substance use in the 12 months prior to screening (including having been hospitalized for such in an in-patient or out-patient intervention program)
* Use of investigational product(s) in another research study within 30 days prior to the baseline visit or during the study duration
* Using any of the following drugs:

  * Antacids or proton pump inhibitors, H2 blockers
  * Salicylates, aspirin, corticosteroids, nonsteroidal anti-inflammatory drugs
  * Anticoagulants, antiplatelet compounds
  * Drugs with known contraindication with iron supplementation or fortification
  * Antiviral medications
  * Levothyroxine (Synthroid)
* Known medical history of specific conditions including:

  * Gastrointestinal disorders: celiac disease, ulcerative colitis, and Crohn's disease
  * Gastric cancer and gastric polyps
  * Colon cancer
  * Diverticular bleeding
  * Inflammatory bowel diseases
  * Angiodysplasia
  * Helicobacter pylori infection
  * Hookworm (Ancylostoma duodenale and Necator americanus)
  * Defects of hemostasis (hereditary hemorrhagic telangectasia, von Willebrand disease)
  * Gastrectomy, duodenal bypass, bariatric surgery
  * Erythropoiesis-stimulating agent therapy
  * Chronic kidney disease
  * Hemochromatosis
  * Hemoglobinopathies
  * Blood clotting disorder
* Have any other active or unstable medical conditions or use of medications/supplements/ therapies that according to the scientific literature, may adversely affect the participant's ability to complete the study or its measures or pose a significant risk to the participant or the quality of the study data.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women
Enrollment: 150 (Estimated)
Dates: Start 2023-04-27 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Serum ferritin (SF) concentrations between active intervention and placebo groups at endline (six months). Proportion of participants remaining iron deficient between active intervention and placebo groups at six months. | Six months
  SF concentrations will be measured using standard clinical lab assay.

SECONDARY OUTCOMES:
Change in SF concentrations from enrolment (baseline), to midline (three months), and endline (six months). | Baseline, three months, six months
  SF concentrations will be measured using standard clinical lab assay.
Change in haemoglobin (Hb) concentrations from enrolment (baseline), to midline (three months), and endline (six months). | Baseline, three months, six months
  Hb concentrations will be measured using standard clinical lab assay.
Levels of metabolites (circulating metabolome) at baseline, three months, and six months. | Baseline, three months, six months
  Functional metabolites in plasma will be measured by Liquid Chromatography-Mass Spectrometry (LC-MS) and Inductively Coupled Plasma-Mass Spectrometry (ICP-MS).
Concentrations of key circulating pro-inflammatory biomarkers at baseline, three months, and six months. | Baseline, three months, six months
  Plasma pro-inflammatory biomarkers will be measured using standard protocols via multi-plex assay (Human Cytokine 27-plex Assay, BioRad) which includes biomarkers such as TNF-alpha, IL-6, MCP-1. The assay will be conducted, and biomarkers measured according to manufacturer's guidelines.
Dietary recall: proportion of participants meeting dietary reference intakes at baseline, three months, and six months. | Baseline, three months, six months
  Mean food and nutrient intakes will be used to determine proportion of participants meeting dietary reference intakes. Dietary recalls will be conducted using the Automated Self-Administered 24-hour Dietary Assessment Tool (ASA24) Canada 2018. This tool measures all food and beverages consumed over a 24-hour period. Dietary recalls will be considered complete if participants provide a minimum of two days of 24-hour recall.
Dietary recall: dietary patterns at baseline, three months, and six months. | Baseline, three months, six months
  Mean food and nutrient intakes will be used to determine dietary patterns of foods known to alter iron absorption.
Dietary recall: Healthy Eating Index (HEI) at baseline, three months, and six months. | Baseline, three months, six months
  Mean food and nutrient intakes will be used to determine HEI scores.
Dietary recall: Dietary Inflammatory Index (DII) at baseline, three months, and six months. | Baseline, three months, six months
  Mean food and nutrient intakes will be used to determine DII scores.
Self-reported perceptions of health at baseline and six months. | Baseline, six months
  Proportion of participants reporting overall good health status will be measured at baseline and at six months. A descriptive health profile will be generated based on health dimensions in both the active intervention and placebo groups. Number of patients, proportions of categorical responses for each health dimensions, including the severity of the health concern will be derived. The investigators will explore significance of change in health profile within each group and significance of the difference between the active intervention and placebo groups at six months. The investigators will assess associations of health profile with adherence to study regimen.
Feasibility: Adherence to the consumption regimen for the regular use of the powder. | Bi-weekly through study completion, approximately 7 months
  Proportion of participants with >80% adherence (defined as preparation and consumption of the powder on at least 4 days per week or a minimum of every second day for the duration of the trial) will be measured bi-weekly for the duration of the trial. Adherence will be determined using the study diary, in which participants will report which days they consumed the study product and which days they did not. Adherence will be reported by participants bi-weekly for the duration of the study.
Feasibility: Adherence to the consumption regimen for the regular use of the powder at three months and six months. | Baseline, three months, six months
  Proportion of unused powder sachets will be measured at three and six months. Participants will be asked to return all used (opened) and unused (unopened) powder sachets at three months and six months. Proportion of unused sachets will be calculated.
Feasibility: Self-reported barriers to use of the powder. | Six months
  Proportion of participants reporting perceived barriers to use of the study product at six months. Qualitative summary of types of perceived barriers at six months.
Palatability. | Six months
  Palatability (i.e. odour, colour, and taste assessments) collected at six months. Palatability assessments of the study product will be conducted at six months using a 9-point hedonic scale to generate palatability scores (where >/=5 indicates that the solution was liked). Differences in participant palatability scores (for colour, odour, sweet, sour, bitter, salty, umami and overall liking) and proportion of participants willing to drink the sample daily will be used to assess the palatability of the powder, show whether the powder is accepted by consumers, and document relationships between palatability and adherence.
Economic: Overall health status. | Six months
  Overall health status will be measured by the EuroQol-5D visual analogue scale (EQ-5D VAS) at six months. The EQ-5D VAS provides a score of 0 to 100, where 0 represents the worst imaginable health status and 100 represents the best imaginable health status.
Economic: Health state/health state index. | Six months
  Health state values will be measure by EuroQol-5D (EQ-5D) at six months. Health state values will be used to generate health state index score using Canadian valuation of EQ-5D health states.
Economic: Quality adjusted life years (QALYs). | Six months
  Health state index scores derived from the EuroQol-5D (EQ-5D) at six months will be used to calculate quality-adjusted life years (QALYs), which will be used to perform cost effectiveness analysis.
Safety (adverse events/harms). | Baseline, three months, six months, and seven months
  Proportion of adverse events (AEs) and proportion of withdrawals from the study due to harms will be measured at baseline, three months, six months, and approximately seven months (four weeks post study end). AE/harms monitoring will occur bi-weekly for the duration of the study and up to four weeks after last study visit for unresolved AEs.

OTHER OUTCOMES:
Exploratory: Microbial metagenome. | Baseline, three months, six months
  The gut microbial metagenome at baseline, three months, and six months. Bacterial genomic DNA will be isolated from stool samples and analysed by whole genome sequencing. Outcomes will be reported descriptively in placebo and intervention groups for: relative abundance, diversity, and variance.
Exploratory: Microbial metagenome inferred function. | Baseline, three months, six months
  Exploratory analyses of inferred function of the metagenome at baseline, three months, and six months. Compositional approaches and Ingenuity Pathway Analysis will be used to generate hypotheses of genes, networks and biological pathways and processes that may be inﬂuenced by the intervention, accounting for clinical data.
Exploratory: Microbial metabolome. | Baseline, three months, six months
  The gut metabolome at baseline, three months, and six months. Microbial metabolome will be measured in placebo and intervention groups and data related to computationally-derived functions from metagenome data) using Liquid Chromatography-Mass Spectrometry (LC-MS) and Inductively Coupled Plasma-Mass Spectrometry (ICP-MS). Data will be processed under standard pipelines with visualisation and pathway analysis by Agilent Mass Proﬁler, MetaboAnalyst and KEGG databases.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Connor, PhD, Principal Investigator — Carleton University; Bénédicte Fontaine-Bisson, RD, PhD, Principal Investigator — University of Ottawa
Locations (1):
- Carleton University, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Subar AF, Kirkpatrick SI, Mittl B, Zimmerman TP, Thompson FE, Bingley C, Willis G, Islam NG, Baranowski T, McNutt S, Potischman N. The Automated Self-Administered 24-hour dietary recall (ASA24): a resource for researchers, clinicians, and educators from the National Cancer Institute. J Acad Nutr Diet. 2012 Aug;112(8):1134-7. doi: 10.1016/j.jand.2012.04.016. Epub 2012 Jun 15. No abstract available. PMID 22704899
- [Background] Bansback N, Tsuchiya A, Brazier J, Anis A. Canadian valuation of EQ-5D health states: preliminary value set and considerations for future valuation studies. PLoS One. 2012;7(2):e31115. doi: 10.1371/journal.pone.0031115. Epub 2012 Feb 6. PMID 22328929
- [Background] Devlin N, Parkin D, Janssen B. Methods for Analysing and Reporting EQ-5D Data [Internet]. Cham (CH): Springer; 2020. No abstract available. Available from http://www.ncbi.nlm.nih.gov/books/NBK565678/ PMID 33347096
- [Background] Gloor GB, Hummelen R, Macklaim JM, Dickson RJ, Fernandes AD, MacPhee R, Reid G. Microbiome profiling by illumina sequencing of combinatorial sequence-tagged PCR products. PLoS One. 2010 Oct 26;5(10):e15406. doi: 10.1371/journal.pone.0015406. PMID 21048977
- [Background] Gloor GB, Wu JR, Pawlowsky-Glahn V, Egozcue JJ. It's all relative: analyzing microbiome data as compositions. Ann Epidemiol. 2016 May;26(5):322-9. doi: 10.1016/j.annepidem.2016.03.003. Epub 2016 Apr 2. PMID 27143475
- [Background] Fernandes AD, Reid JN, Macklaim JM, McMurrough TA, Edgell DR, Gloor GB. Unifying the analysis of high-throughput sequencing datasets: characterizing RNA-seq, 16S rRNA gene sequencing and selective growth experiments by compositional data analysis. Microbiome. 2014 May 5;2:15. doi: 10.1186/2049-2618-2-15. eCollection 2014. PMID 24910773
- [Background] Zierer J, Jackson MA, Kastenmuller G, Mangino M, Long T, Telenti A, Mohney RP, Small KS, Bell JT, Steves CJ, Valdes AM, Spector TD, Menni C. The fecal metabolome as a functional readout of the gut microbiome. Nat Genet. 2018 Jun;50(6):790-795. doi: 10.1038/s41588-018-0135-7. Epub 2018 May 28. PMID 29808030
- [Background] Abdel Rahman AM, Pawling J, Ryczko M, Caudy AA, Dennis JW. Targeted metabolomics in cultured cells and tissues by mass spectrometry: method development and validation. Anal Chim Acta. 2014 Oct 3;845:53-61. doi: 10.1016/j.aca.2014.06.012. Epub 2014 Jun 12. PMID 25201272